CLINICAL TRIAL: NCT06631053
Title: Use of Velocity Monitoring to Prescribe Appropriate Flywheel-based Inertial Training (FIT) Workloads for Exercise in Space Flight
Brief Title: FIT Exercise in 30d of ULLS-induced Muscle Disuse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lance Bollinger (Other)
Collaborators: University of Louisville (Other); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lance Bollinger, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97289; 80NSSC24M0149 (Other Grant/Funding Number: NASA)
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Muscle Atrophy; Muscle Weakness
Keywords: spaceflight; unweighting; disuse; exercise
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness; Motor Activity

STUDY DESIGN:
Intervention Model Description: ULLS is the gold standard for assessing muscle disuse in ambulatory subjects. Velocity based resistance training and High Intensity Interval Training are gold-standard exercise strategies in terrestrial settings which tend to out-perform other exercise interventions. However, these exercise paradigms have not be applied to those undergoing unloading such as astronauts in space flight. Here, we aim to adopt principles from these established exercise interventions to determine their effectiveness in preserving muscle and aerobic fitness during 30d ULLS.
Masking Description: Participants are unable to be masked to their intervention (exercise v. non-exercise). Although other researchers from this team will be responsible for directly implementing exercise interventions, exercise sessions will be conducted in the same building as the PI's office. Therefore, it is likely that the PI will be aware of which subjects are completing exercise sessions. The PI and his team will be directly responsible for assessing primary and secondary research outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Exercise (Active Comparator): Participants will undergo a 30d Unilateral Lower Limb Suspension (ULLS) without exercise
  Interventions: Other: No Exercise
- velocity-based FIT (VBFIT) (Experimental): Participants will undergo a 30d Unilateral Lower Limb Suspension (ULLS) with exercise
  Interventions: Other: velocity-based FIT (VBFIT)

INTERVENTIONS:
Other: velocity-based FIT (VBFIT) — Participants will ambulate unilaterally using a shoe modified with a 5cm rocker-style stack and forearm crutches for the duration of the study.
  All participants will complete two testing sessions prior to ULLS, one testing session at day 13, and two testing sessions at the end of the study. Those assigned to the exercise group will perform a both high-intensity resistance and aerobic exercise three times per week
  Arms: velocity-based FIT (VBFIT)
Other: No Exercise — Participants will ambulate unilaterally using a shoe modified with a 5cm rocker-style stack and forearm crutches for the duration of the study.
  All participants will complete two testing sessions prior to ULLS, one testing session at day 13, and two testing sessions at the end of the study.
  Arms: No Exercise

SUMMARY:
This study aims to determine how flywheel-based inertial training (FIT) implemented according to principles of velocity-based training (VBT) and High-Intensity Interval Training (HIIT) affects disuse-induced physical de-conditioning including loss of voluntary muscle strength, aerobic capacity, and balance regulation.

DETAILED DESCRIPTION:
The primary objectives of this project are:

1. To assess how 30d of unilateral lower limb suspension (ULLS) with and without FIT exercise affects voluntary and electrically-evoked twitch force, motor unit recruitment, and anisotropic measures.
2. To determine how muscle anisotropy (assessed through diffusion tensor imaging) and motor unit action potential train (MUAPT) characteristics relate to contractile function in loaded and unloaded limbs

Secondary objectives include:

1. To assess impact of ULLS with and without FIT on aerobic capacity
2. To assess impact of ULLS with and without FIT on balance regulation during single-leg stance

This study aims to recruit 10 healthy, physically active participants (both male and female). Participants will undergo 30d of ULLS to unload the left limb during daily living activities. Subjects will wear a specially modified shoe with a 5cm rocker-style stack on the right leg and ambulate using crutches. Participants will be randomly assigned to either a control or exercise group. Those in the exercise group will perform Flywheel-based Inertial Training (FIT) leg press three times per week. Moment of inertia of the flywheel will be adjusted to elicit movement speeds of 0.4 m/s for resistance training (four sets of 10 repetitions). For High Intensity Interval Training, flywheel moment of inertia will be adjusted to elicit movement speed of 1.0m/s during upright squats (four sets of 3 min).

Before and after the intervention, subjects will complete a series of tests including:

1. Body Composition - height, weight, waist circumference, and tetrapolar bioelectrical impedance analysis will be conducted.
2. Balance assessment - center of pressure will be assessed using portable force decks during single leg stance with eyes open and closed. This test will be repeated in the shod and unshod conditions. MUAPT data (high density surface electromyography) will be collected for the soleus and tibialis anterior during this test.
3. Aerobic capacity test - VO2max will be determined during a graded exercise test on a cycle ergometer (3 min per stage). Gas exchange and heart rate data will be collected continuously throughout the test. Pedal force will also be assessed. Additional outcomes such as ventilatory threshold and substrate utilization will be assessed.
4. Muscle Imaging - Diffusion tensor imaging (DTI), a magnetic resonance technique will be used to assess anisotropic measures, muscle volume, fascicle length, and fascicle orientation of the mid-thigh.
5. Muscle strength testing - Maximal voluntary isometric and isokinetic strength of the knee extensors, flexors, and ankle plantar- and dorsi-flexors will be assessed. Interpolated twitch (electrical stimulation of the femoral nerve) will be used to assess twitch characteristics and voluntary activation of the quadriceps

ELIGIBILITY:
Inclusion Criteria:

* Regularly engaging in aerobic exercise (> 150min/wk) and resistance exercise (>1 time per week) for the past 12 months
* Education greater than or equal to bachelor's degree (any field)

Exclusion Criteria:

* Waist circumference < 55cm or > 90cm (F) and < 75cm or > 100cm (M)
* Body mass index < 18.5 or > 29.9
* Shoe size < 25 or >29cm.
* Not regularly engaging in exercise for previous 12 months
* Tobacco use within previous 6 months
* Blood clotting disorder
* Heart arrhythmia
* Implanted device which could negatively be affected by electrical impulse or strong magnetic field such as pacemaker, internal defibrillator, or cochlear implant
* Diagnosed cardiovascular, pulmonary, renal, or metabolic disease
* Pregnancy (within previous 6 months)
* Oral contraceptive use (within previous three months)
* High resting blood pressure (>140 systolic and/or > 90 diastolic)
* Currently or previously undergone gender-affirming therapy (hormone therapy or sexual reassignment surgery)
* Low back or leg injury in previous 6 months
* Currently taking medication to assist with sleep
* Muscle, bone, or joint injury that limits physical activity within previous 6 months
* Neurological disorder which affects balance (such as multiple sclerosis or Parkinson's disease)

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Voluntary activation | Baseline, day 13, and day 30
  Voluntary activation of the quadriceps will be assessed with electrical stimulation of the femoral nerve before, during, and after a maximal voluntary isometric contraction (MVIC) using the interpolated twitch technique.
Twitch Properties-Electromechanical Delay | Baseline, day 13, and day 30
  Electromechanical delay will be calculated as the time difference between the onset of electrical impulse and onset of torque development during femoral nerve stimulation. This will be measured before and after a maximal voluntary isometric contraction.
Twitch Properties-Rate of Torque Development | Baseline, day 13, and day 30
  Rate of Torque Development will be calculated as the change in torque divided by the change in time in the linear phase between 20 and 80% of peak twitch torque during femoral nerve stimulation. This will be measured before and after a maximal voluntary isometric contraction.
Twitch Properties-Time to peak Tension | Baseline, day 13, and day 30
  Time to peak tension will be calculated as the time difference between the onset of electrical impulse and peak twitch torque during femoral nerve stimulation. This will be measured before and after a maximal voluntary isometric contraction.
Twitch Properties-Peak Twitch Torque | Baseline, day 13, and day 30
  Peak twitch torque during femoral nerve stimulation will be calculated as the highest torque output immediately (approximately 200ms) following femoral nerve stimulation. This will be measured before and after a maximal voluntary isometric contraction.
Twitch Properties-Relaxation Rate | Baseline, day 13, and day 30
  Relaxation rate will be calculated as the change in torque divided by the change in time during the relaxation phase of twitch following femoral nerve stimulation. This will be measured before and after a maximal voluntary isometric contraction.
Post activation Potentiation | Baseline, day 13, and day 30
  Post-activation will be calculated as the percentage difference in peak twitch torque in femoral nerve stimulation before and after a maximal voluntary isometric contraction.
Motor unit action potential train (MUAPT) firing rate | Baseline, day 13, and day 30
  Firing rate of individual motor units of the vastus lateralis (VL) will be assessed with high density surface electromyography (EMG) using four-pin high density surface electromyography electrodes. Firing rate at 30, 60, and 90% MVIC will be reported. Motor unit firing rate will also be reported during static stance.
  Participants will use a screen displaying real-time torque output. Participants will voluntarily increase torque (5 seconds), hold at a pre-determined torque level (10 seconds), and gradually reduce force back to resting (5 seconds) with the knee held in a fixed position. This test will be completed with a 10s isometric hold at 30, 60, and 90% of maximal voluntary isometric force.
Motor unit action potential train (MUAPT) recruitment threshold. | Baseline, day 13, and day 30
  Recruitment threshold of individual motor units of the VL will be assessed with high density surface electromyography using four-pin high density surface electromyography electrodes. Recruitment threshold will be measured during isometric ramp contractions of the quadriceps
  Participants will use a screen displaying real-time torque output. Participants will voluntarily increase torque (5 seconds), hold at a pre-determined torque level (10 seconds), and gradually reduce force back to resting (5 seconds) with the knee held in a fixed position. This test will be completed with a 10s isometric hold at 30, 60, and 90% of maximal voluntary isometric force.
Motor unit action potential train (MUAPT) de-recruitment threshold. | Baseline, day 13, and day 30
  De-recruitment threshold of individual motor units f the VL will be assessed with high density surface electromyography using four-pin high density surface electromyography electrodes. Recruitment threshold will be measured during isometric ramp contractions of the quadriceps
  Participants will use a screen displaying real-time torque output. Participants will voluntarily increase torque (5 seconds), hold at a pre-determined torque level (10 seconds), and gradually reduce force back to resting (5 seconds) with the knee held in a fixed position. This test will be completed with a 10s isometric hold at 30, 60, and 90% of maximal voluntary isometric force.
Muscle size | Baseline and day 30
  Muscle size will be measured by MRI. Anatomical MRI scans will allow for assessment of anatomical cross sectional area.
Muscle Physiological cross-sectional area | Baseline and day 30
  Diffusion tensor imaging (DTI) will be used to assess muscle volume and fascicle length. Physiological cross-sectional area will be calculated as Muscle volume divided by fascicle length.
Muscle Fractional Anisotropy | Baseline and day 30
  Diffusion tensor imaging (DTI) will be used to assess anisotropic measures. A ratio of the diffusivity in the principal planes will be used to calculate fractional anisotropy.
Muscle Diffusion properties | Baseline and day 30
  Diffusion tensor imaging (DTI) will be used to assess rate of water diffusion in three principal planes. We will report rates of water diffusion in three ways: 1) mean diffusivity (average rate in all three plane), 2) axial diffusivity (rate of diffusion along primary axis), and 3) radial diffusivity (rate of diffusion perpendicular to the primary axis).
Muscle cross-sectional area (Ultrasound) | Baseline, day 13, and day 30
  cross-sectional area of the vastus lateralis and rectus femoris will be measured by ultrasonography
Fascicle length | Baseline, day 13, and day 30
  Panoramic views of the mid-portion of the VL will be measured by ultrasonography
Pennation angle | Baseline, day 13, and day 30
  Pennation angle of the mid-portion of the vastus lateralis will be assessed by ultrasonography
Voluntary Isokinetic Muscle Strength | Baseline, day 13, and day 30
  Maximal voluntary isokinetic concentric strength of the knee extensors/flexors and ankle dorsi-/plantar-flexors will be assessed at 60 deg/s
Voluntary Isometric Muscle Strength | Baseline, day 13, and day 30
  Maximal voluntary isometric strength of the knee extensors/flexors and ankle dorsi-/plantar-flexors will be assessed during a (10 seconds) maximal effort contraction.

SECONDARY OUTCOMES:
Aerobic Capacity | Baseline and day 30
  Subjects will complete a VO2max exercise test on a stationary bicycle. Gas exchange and heart rate data will be collected continuously. Initial workload will be set at approximately 2 METS. Every three minutes, we will add more resistance to the pedals (~1.5 METS). Subjects will continue to pedal until they can either not maintain pedal speed (50RPM) or until a plateau in VO2 occurs. Pedal force for each limb will be assessed.
Ventilatory Threshold | Baseline and day 30
  Gas exchange data from the aerobic capacity test (VO2, ventilation; VE, and VCO2) will be used to calculate ventilatory threshold during exercise
Substrate utilization | Baseline and day 30
  Gas exchange data from the aerobic capacity test (VO2, respiratory exchange ratio; RER, and VCO2) will be used to calculate substrate utilization (energy expenditure, carbohydrate use, and fatty acid oxidation) at varying exercise intensities
Body Composition | Baseline and day 30
  Bioelectrical Impedance Analysis (BIA) will be used to assess body composition. Subjects will lie supine and have small adhesive electrodes placed on the right hand, wrist, ankle, and foot. A small (imperceptible) electrical current will be delivered to one electrode and the amount of resistance to the electrical current will be used to measure body composition. Percent body fat will be measured. Muscle mass will be calculated using previously established formulae.
Postural sway area | Baseline, day 13, and day 30
  Subjects will complete a series of balance assessments while standing on one leg using a dual force plate system. Subjects will stand still on one leg for 15 seconds with hands on hips. This will be repeated on both legs with eyes open and with eyes closed in the shod and unshod conditions in random order. Postural sway area will be calculated as an index of postural control.
Postural Sway Velocity | Baseline, day 13, and day 30
  Subjects will complete a series of balance assessments while standing on one leg using a dual force plate system. Subjects will stand still on one leg for 15 seconds with hands on hips. This will be repeated on both legs with eyes open and with eyes closed in the shod and unshod conditions in random order. Mean Postural sway velocity will be calculated as an index of postural control.
Motor unit firing rate - single leg stance | Baseline, day 13, and day 30
  Subjects will complete a series of balance assessments while standing on one leg using a dual force plate system. Subjects will stand still on one leg for 15 seconds with hands on hips. This will be repeated on both legs with eyes open and with eyes closed in the shod and unshod conditions in random order.
  High density surface EMG sensors will be adhered to the skin over the tibialis anterior and soleus muscles with double-sided tape. Exponential functions will be fit to describe the relationship between motor unit firing rate and action potential amplitude on an individual manner to determine how firing rates of various motor unit pools relate to postural control.
Change in heart rate at rest | Baseline and day 30
  heart rate measured
Change in blood pressure at rest | Baseline and day 30
  blood pressure measured at the arm
Change in heart rate variability | Baseline and day 30
  for 20 minutes electrodes will be placed on the skin of the chest and a respiratory belt will be wrapped around the chest and blood pressure will be taken at the arm. During the final 10 minutes, 5 minutes of regular breathing (minutes 11-15), and 5 minutes of controlled breathing at a rate of 12 breaths per minute will be done. Resting heart rate (throughout), respiratory rate (throughout) and blood pressure (min 15 and 20) will be collected.
Change in heart rate recovery after exercise | Baseline and day 30
  a maximal-effort exercise test on a stationary bicycle will be done. Immediately upon finishing the cycling, participants will rest on the bike for 5 minutes while remaining as still as possible. Heart rate will be collected throughout the this time to give a measure of heart rate recovery

CONTACTS AND LOCATIONS:
Overall Officials: Lance Bollinger, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No